CLINICAL TRIAL: NCT04581252
Title: Heart Failure HemOdynamic Prognostic Evaluation and OutcomE (HF-HOPE) Study
Acronym: HF-HOPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ashish H Shah, Assistant Professor, University of Manitoba
Other Study IDs: HS23206
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non-invasive cardiac system — Non-invasive cardiac system

SUMMARY:
Summary of the HF-HOPE study:

Background and existing knowledge gap:

As per the Canadian Chronic Disease Surveillance System, about 1 in 12 Canadian adults aged ≥20 live with diagnosed heart disease. Every hour, about 12 Canadian adults aged ≥20 die due to heart failure (HF). It is estimated that HF results in direct costs of more than $2.8 billion per year in Canada alone. As per the Canadian Society of Cardiology, heart failure is defined as "a complex clinical syndrome in which abnormal heart function results in, or increases the subsequent risk of, clinical symptoms and signs of reduced cardiac output and/or pulmonary or systemic congestion at rest or with stress". Although HF is defined as "reduced cardiac output state" no objective parameters are set to define the condition. Invasive monitoring is routinely used in hemodynamic evaluation of critically ill patients admitted in the hospital, however, there is no reliable tool available to measure hemodynamic parameters that may predict, immediate or long-term, risk of worst health outcomes in stable HF patients. We hypothesize that non-invasive bioimpedance-based hemodynamic parameters can be used as a predictive tool for health outcomes in patients with HF. To ascertain this, we propose the first of its kind HF-HOPE study.

Objectives of HF-HOPE study are to 1) characterize hemodynamic measures of resting versus post-exercise (mounted ergometer) in patients with all-comer stable HF subjects, irrespective of their HF etiology using Non-Invasive Cardiac System (NICaS); 2) correlate NICaS-derived hemodynamic parameters to identify, early- and long-term risk of worse health outcomes (unplanned hospital admission due to HF or arrhythmias; listing for heart transplantation/palliative care; and death); 3) correlate the lean body mass (muscle and skeleton) with their body mass index (kg/m2) and the risk of worse health outcomes; and 4) Nested cohort study: identify the outcome-associated biomarkers of chronic HF by employing a non-targeted metabolomics/lipidomics approach.

Methods: The HF-HOPE is a single center, prospective, double-blind, pragmatic clinical study. It will be conducted at St. Boniface general hospital, Manitoba's tertiary cardiac center. Patients aged ≥18 years, irrespective of any sex or gender, with confirmed diagnosis of HF will be enrolled in the study. Hemodynamic measurements (stroke volume, cardiac output, cardiac index, total peripheral vascular resistance, and cardiac power index) will be assessed using NICaS at 3-times (at rest in supine, siting position as well as after exercise on a mounted ergometer) at baseline and 6 months (±1 month) in each enrolled participant. Patients will be followed to record health outcomes as outlined above, each year. The BodPod, air displacement plathysmography device will be used to determine body compositions at baseline and 6-month. Baseline demographic data will be gathered. To optimize the use of clinical resources, we will collect blood and urine samples for non-selective metabolomics and lipidomics profiling by adopting -omics approach as a nested cohort study. Statistical analysis: Assuming the 8 to 12% 1-year mortality rate following admission with HF, a projected sample size of 500 would be suffice. Conservatively 4 covariates will be included in multivariable statistical models, while testing the independent effect of the relevant NICaS parameters of interest. We will perform subgroup analysis using age, sex, ethnicity, concomitant disease conditions, medications, and lean body mass.

Anticipated outcomes and future implications: The HF-HOPE study is the first of its kind study employing non-invasive hemodynamic parameters to predict worsening health outcomes over time in HF patients. The successful outcomes will provide a promising cost effective, rapid, and reliable tool to predict worsening health outcomes before it actually lead to hospitalization, tissue damage or death. This early warnings will provide adequate time for appropriate intervention. The HF- HOPE study has been meticulously designed to replicate the pragmatic conditions while assessing the non-invasive hemodynamic measurements to widen the knowledge translation of outcomes to change the clinical practice of HF patient management. Further, this may provide supporting data for future randomized trial to replace the costly, resource-intense, and complex invasive tool to determine hemodynamic measurements in HF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age with the confirmed diagnosis of HF with a stable condition over last 3 months, irrespective of underlying etiology and time of index diagnosis (> 3 months).
2. Should be able to understand and willing to sign the consent form.

Exclusion Criteria:

1. Recent worsening of clinical state (increase dose of diuretics or unplanned hospital admission due to HF or arrhythmia over the last 3 months)
2. Cancer or terminal illness that may adversely affect lifespan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
the composite score of 1) recurrent hospital admission due to HF or arrhythmias, 2) heart transplantation/palliative care, and 3) death | 1 year
  Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Result] Ezekowitz JA, O'Meara E, McDonald MA, Abrams H, Chan M, Ducharme A, Giannetti N, Grzeslo A, Hamilton PG, Heckman GA, Howlett JG, Koshman SL, Lepage S, McKelvie RS, Moe GW, Rajda M, Swiggum E, Virani SA, Zieroth S, Al-Hesayen A, Cohen-Solal A, D'Astous M, De S, Estrella-Holder E, Fremes S, Green L, Haddad H, Harkness K, Hernandez AF, Kouz S, LeBlanc MH, Masoudi FA, Ross HJ, Roussin A, Sussex B. 2017 Comprehensive Update of the Canadian Cardiovascular Society Guidelines for the Management of Heart Failure. Can J Cardiol. 2017 Nov;33(11):1342-1433. doi: 10.1016/j.cjca.2017.08.022. Epub 2017 Sep 6. PMID 29111106
- [Result] Chomsky DB, Lang CC, Rayos GH, Shyr Y, Yeoh TK, Pierson RN 3rd, Davis SF, Wilson JR. Hemodynamic exercise testing. A valuable tool in the selection of cardiac transplantation candidates. Circulation. 1996 Dec 15;94(12):3176-83. doi: 10.1161/01.cir.94.12.3176. PMID 8989126
- [Result] Lee DH, Keum N, Hu FB, Orav EJ, Rimm EB, Willett WC, Giovannucci EL. Predicted lean body mass, fat mass, and all cause and cause specific mortality in men: prospective US cohort study. BMJ. 2018 Jul 3;362:k2575. doi: 10.1136/bmj.k2575. PMID 29970408